CLINICAL TRIAL: NCT03597061
Title: Healthy Start to Feeding Pilot Trial
Brief Title: Healthy Start to Feeding Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Cathy Stough, Assistant Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-7248
Record Dates: First submitted 2018-06-27; First posted 2018-07-24 (Actual); Results first posted 2021-07-15 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Weight, Body; Diet Habit
Keywords: obesity prevention; infant; complementary feeding; diet variety; weight-for-length; food responsiveness; satiety responsiveness
MeSH Terms: conditions — Body Weight; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Infants will be assigned to either the treatment or control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Start to Feeding Intervention (Experimental): Participants and their parents will participate in a 3 session intervention targeting healthy introduction of complementary foods. Intervention sessions will occur when the infant is 4, 6, and 9 months of age.
  Interventions: Behavioral: Healthy Start to Feeding
- Control (No Intervention): Participants and their parents will complete pre- and post-treatment period study visits to assess study outcomes. They will receive no intervention.

INTERVENTIONS:
Behavioral: Healthy Start to Feeding — The intervention provides parent education and skills training on a responsive feeding approach to introduction of healthy foods in infancy. Session content is manualized and administered by interventionists with expertise in child development and behavioral strategies for managing child eating behaviors under the supervision of a licensed clinical child psychologist and pediatric occupational therapist. Sessions are conducted individually with participants and primary caregivers and include educational content, handouts and instructions, modeling of skills by the interventionist, caregiver practicing of skills in session, establishment of behavioral goals, and problem solving barriers to implementation of treatment content. Content will include topics such as allowing infants' own hunger and satiety cues to guide the feeding experience, introducing healthy foods, parental attunement to infant satiety cues, and promoting infants' own self-feeding.
  Arms: Healthy Start to Feeding Intervention

SUMMARY:
The current study will test the impact of a 3-session obesity prevention program targeting healthy introduction of solid foods in infancy on growth trajectories, appetite regulation, and diet. The investigators will also test the feasibility and family satisfaction with the treatment. Healthy infants with normal and elevated weight-for-length will be enrolled in the study at 3 months of age and complete an initial study visit to assess baseline anthropometrics,demographics, parental feeding practices and beliefs, and infant appetite. Infants will than be randomly assigned to either the treatment condition (n = 20) or control condition (n = 20). Infants in the control condition will receive no intervention or further contact with the study team besides for completion of a final study assessment visit when the child is 9 months old. Infants in the treatment condition will receive a 3 session intervention targeting healthy introduction of solid foods, with study visits occurring when the child is 4 months, 6 months, and 9 months old. All families will complete a final study visit to complete post-treatment period measurements, which will include infant anthropometrics and parent-report of infant appetite, infant diet, and parental feeding practices and beliefs. Outcomes include: weight-for-length percentile, infant satiety responsiveness, infant food responsiveness, and infant fruit and vegetable consumption. Family satisfaction and treatment attendance will also be assessed.

DETAILED DESCRIPTION:
The purpose of this research study is to pilot test a prevention program to promote healthy introduction of solid foods and healthy weight gain among infants. Introduction of complementary foods (i.e., foods besides formula or breast milk) represents a major dietary milestone for infants. The current study will test the feasibility of a 3-session intervention encouraging healthy introduction of complementary foods and use of a responsive feeding approach. Feasibility of the intervention and the impact of the Healthy Start to Feeding (HSF) intervention on obesity risk factors and growth will be explored. This will be achieved through exploration of the following aims and hypotheses:

Aim 1: Determine feasibility of the intervention and family satisfaction with the treatment.

H1: Families assigned to the intervention condition will attend equal to or greater than 67% of treatment sessions.

H2: Families receiving the intervention will rate the program as helpful and consistent with the families' needs and priorities.

Aim 2: Test the impact of the HSF intervention on growth trajectories, appetite regulation, and diet at post-treatment.

H1: Infants receiving the intervention will experience lower incidence of high weight-for-length (> 85th percentile) compared to infants in the control condition.

H2: Infants in the treatment condition will show greater satiety responsiveness and lower food responsiveness as assessed through a well-validated parent-report measure (Baby Eating Behavior Questionnaire; Llewellyn, van Jaarsveld, Johnson, Carnell, & Wardle, 2010).

H3: Infants in the treatment condition will consume a greater variety of fruits and vegetables than infants in the control condition as assessed through a food frequency questionnaire completed by parents.

ELIGIBILITY:
Inclusion Criteria:

* Infant aged 2-3 months at study recruitment
* Infant not previously introduced to complementary foods (i.e., any food besides formula or breastmilk)
* Infant born at > 38 weeks gestation
* Infant weight-for-length > 10th percentile
* Parent is fluent English speaker

Exclusion Criteria:

* Known infant developmental delay
* Impaired infant fine or gross motor skills
* Condition currently impacting the infant's feeding and eating

Ages: 3 Months to 10 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathleen Stough, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected will be shared through 1) dissemination of aggregate data through scientific publication, summary on the research laboratory's website, and presentation at regional, national, and international conferences and 2) availability of data to requesting researchers and investigators. Researchers interested in receiving the dataset should request the dataset from the principal investigator.
  In addition to these two avenues for data sharing, if provided the opportunity at the time of publication, the dataset will be uploaded to any data repository offered through the scientific journal in which findings are published.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data collected at baseline will be made available at the time of acceptance of the first publication presenting this data, which will be submitted for publication no later than 1 year following the completion of baseline data collection. All other data collected throughout the project will be made available at the time of acceptance of the primary treatment outcomes paper, which will be submitted for publication no later than 1 year following the completion of the last post-treatment visit.
Access Criteria: Requesting researchers and investigators will be asked to use the data only for IRB-approved or exempted research purposes and to present only aggregate descriptions of data that do not identify any one participant.

REFERENCES:
- [Derived] Ojha S, Elfzzani Z, Kwok TC, Dorling J. Education of family members to support weaning to solids and nutrition in later infancy in term-born infants. Cochrane Database Syst Rev. 2020 Jul 25;7(7):CD012241. doi: 10.1002/14651858.CD012241.pub2. PMID 32710657

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Healthy Start to Feeding Intervention
Started | 17 | 17
Completed | 16 | 16
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Healthy Start to Feeding Intervention: Participants and their parents participated in a 3-session intervention targeting healthy introduction of complementary foods. Intervention sessions occurred when the infant was 4, 6, and 9 months of age.
  Healthy Start to Feeding: The intervention provided parent education and skills training on a responsive feeding approach to introduction of healthy foods in infancy. Session content was manualized and administered by interventionists with expertise in child development and behavioral strategies for managing child eating behaviors under the supervision of a licensed clinical child psychologist and pediatric occupational therapist. Sessions were conducted individually with participants and primary caregivers and included educational content, handouts and instructions, modeling of skills by the interventionist, caregiver practicing of skills in session, establishment of behavioral goals, and problem solving barriers to implementation of treatment content. Content included topics such as allowing infants' own hunger and satiety cues to guide the feeding experience, introducing healthy foods, parental attunement to infant satiety cues, and promoting infants' own self-feeding.
- Control: Participants and their parents completed pre- and post-treatment study visits to assess study outcomes. They received no intervention.
- Total: Total of all reporting groups
Arm/Group | Healthy Start to Feeding Intervention | Control | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 17 | 34
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 16 | 17 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 14 | 30
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Weight-for-Length Percentile
Description: Infant anthropometrics of weight and length were measured and used to calculate weight-for-length percentile standardized for age and gender.
Time Frame: Weight and length were measured at both pre-treatment (when infant was 3 months of age) and post-treatment (when infant was 9 months of age).
Measure: Mean (Standard Deviation); unit: Percentile
Arm/Group | Healthy Start to Feeding Intervention | Control
Number analyzed (Participants) | 16 | 16
Percentile
  Pre-treatment | 44.94 (30.25) | 46.70 (26.97)
  Post-treatment | 58.69 (31.78) | 48.54 (30.82)

2. Primary Outcome: Appetite Regulation
Description: Infant satiety and food responsiveness was measured using the parent-report Baby Eating Behavior Questionnaire (BEBQ). The BEBQ provides subscale scores for "Food Responsiveness", "Enjoyment of Food", "Satiety Responsiveness", and "Slowness in Eating" with each subscale score ranging from 1 to 5, with 5 representing higher values on that construct. Each subscale score is computed as the average of all individual items on that subscales.
Time Frame: The BEBQ was completed at both pre-treatment (when infant is 3 months of age) and post-treatment (when infant is 9 months of age).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Healthy Start to Feeding Intervention | Control
Number analyzed (Participants) | 16 | 16
Score on a scale
  Pre-treatment: Food Responsiveness | 2.96 (.33) | 3.01 (.24)
  Pre-treatment: Enjoyment of Food | 3.61 (.27) | 3.72 (.35)
  Pre-treatment: Satiety Responsiveness | 1.92 (.49) | 1.85 (.30)
  Pre-treatment: Slowness in Eating | 2.59 (.48) | 2.73 (.48)
  Post-treatment: Food Responsiveness | 2.82 (.46) | 2.97 (.29)
  Post-treatment: Enjoyment of Food | 3.70 (.26) | 3.58 (.24)
  Post-treatment: Satiety Responsiveness | 1.54 (.45) | 1.96 (.36)
  Post-treatment: Slowness in Eating | 2.41 (.41) | 2.58 (.35)

3. Primary Outcome: Fruit and Vegetable Variety
Description: Fruit and vegetable variety was assessed using the parent-report Block Food Frequency Questionnaire. Scores were calculated for servings of vegetables per day and servings of fruits per day. The minimum value is 0. There is no upper-bound for the maximum value, as this is dependent on the individual participant's food consumption. Higher numbers indicate greater consumption. Only post-treatment results are presented since infants had not been introduced to solid foods at the time of baseline.
Time Frame: The Block Food Frequency Questionnaire was completed at both pre-treatment (when infant is 3 months of age) and post-treatment (when infant is 9 months of age).
Measure: Mean (Standard Deviation); unit: Servings per day
Arm/Group | Healthy Start to Feeding Intervention | Control
Number analyzed (Participants) | 16 | 16
Servings per day
  Post-treatment: Fruit Servings Per Day | 1.86 (1.19) | 2.19 (1.11)
  Post-treatment: Veggie Servings Per Day | 4.92 (3.63) | 5.10 (3.75)

4. Secondary Outcome: Family Satisfaction - Defined as Appropriateness of the Intervention Content and Session Timing, Clarity of Information, Knowledge of the Recommendations, Helpfulness, and Whether They Would Recommend the Intervention to Others.
Description: Caregivers in the treatment condition completed a survey measuring whether parents found the intervention appropriate for their infant, whether sessions occurred at the right time, whether information was presented clearly, whether they knew how to implement the recommendations, whether the intervention was helpful, whether they were satisfied with the intervention, and whether they would recommend the intervention to a friend/family member/coworker. Each satisfaction attribute will be assessed on a 1-5 Likert scale with higher scores indicating higher agreement. Information from each individual item will be used, and no total or subscale scores will be computed. Parents also provided qualitative information on what additional information should be included in the intervention, what information was not helpful, what should be changed about the intervention, and what should stay the same about the intervention.
Time Frame: The measure of family satisfaction will be completed at post-treatment (when the child is 9 months of age).
Measure: Mean (Standard Deviation); unit: Item scores
Arm/Group | Healthy Start to Feeding Intervention
Number analyzed (Participants) | 15
Item scores
  Appropriateness | 4.60 (1.06)
  Timing | 4.47 (1.13)
  Clarity | 4.67 (1.05)
  Implementation | 4.67 (1.05)
  Helpful | 4.53 (.83)
  Satisfication | 4.47 (1.25)
  Would Recommend | 4.47 (1.19)

5. Secondary Outcome: Treatment Attendance
Description: Treatment attendance was tracked for each family.
Time Frame: Attendance of sessions at study month 2 (session 1), study month 4 (session 2), and study month 7 (session 3) was recorded. The number of sessions that each participant attended was calculated.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Start to Feeding Intervention
Number analyzed (Participants) | 16
Participants
  Attended Session 1 | 16
  Attended Session 2 | 16
  Attended Session 3 | 16

ADVERSE EVENTS:
Time Frame: From baseline to post-treatment (approximately 6 months)
Arm/Group | Healthy Start to Feeding Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/61/NCT03597061/Prot_004.pdf
  • Statistical Analysis Plan (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/61/NCT03597061/SAP_005.pdf
  • Informed Consent Form (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/61/NCT03597061/ICF_006.pdf